CLINICAL TRIAL: NCT03354403
Title: Mothers' Experiences With X-linked Retinoschisis Compared to Fathers' Experiences
Brief Title: Mothers Experiences With X-linked Retinoschisis Compared to Fathers Experiences
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180016; 18-EI-0016
Record Dates: First submitted 2017-11-25; First posted 2017-11-28 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Retinoschisis; X-Linked
Keywords: XLRS; RS1; Carrier
MeSH Terms: conditions — Retinoschisis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Patients: Up to 50 mothers of sons of all ages diagnosed with XLRS are eligible to participate in this study. Up to 50 fathers of sons of all ages with XLRS are also eligible to participate and will serve as a comparison group.

SUMMARY:
Background:

X-linked retinoschisis (XLRS) is a genetic condition. It usually presents in boys in childhood with vision loss. Genetic conditions affect the people who have it and also their family members. Researchers want to learn if mothers and fathers react differently when a son gets XLRS. They also want to learn how personality impacts the way people react. This will help researchers find better ways to support families living with XLRS.

Objective:

To learn more about the experiences of mothers of sons with XLRS compared to fathers of sons with XLRS. Also to study personality differences between mothers and fathers.

Eligibility:

Parents of a biological son of any age with XLRS who is enrolled in protocol 03-EI-0033

Design:

Participants will be asked questions in person or by phone. This will last 30 90 minutes. They will be asked about their experience with XLRS and how it has impacted their family. The interview will be recorded.

Participants will complete a survey about personality traits. It will be anonymous. It can be completed by mail, email, or fax. It will take about 15 minutes.

Participants data may be shared with others, including those not at NIH, if they agree. Their data may be stored.

Sponsoring Institution: National Eye Institute

DETAILED DESCRIPTION:
OBJECTIVE: The objective of this study is to explore the experiences of mothers of sons with X-linked retinoschisis (XLRS) compared to fathers of sons with XLRS and to draft a personality profile of both mothers and fathers based on the findings.

<TAB>

STUDY POPULATION: Up to 50 mothers of sons of all ages diagnosed with XLRS are eligible to participate in this study. Up to 50 fathers of sons of all ages with XLRS are also eligible to participate and will serve as a comparison group.

DESIGN: This is a pilot mixed-methods study that involves a cross sectional qualitative interview and a self-administered questionnaire. Participants will be recruited through a "parent" study "Clinical and Molecular Studies of X-linked Retinoschisis" (03-EI-0033). Interviews will be conducted either in person at the National Institutes of Health Clinical Center (NIH CC) or by telephone. The interview will explore the experiences and impact of having a son with XLRS. Interviews will be recorded, transcribed verbatim, coded by two independent coders, and analyzed thematically. Participants will also be asked to complete a questionnaire to assess personality traits, anxiety, and optimism, using scales shown to be valid and reliable in the general population and in clinical samples. Results from these scales will provide information about variables that cannot be reliably assessed from an interview. This study is not designed to assess causality; rather, it will be used to generate hypotheses and inform future social and behavioral and/or basic science research studies of parents of sons with XLRS.

OUTCOME MEASURES: The primary outcomes of this study include a description of the experiences of mothers of sons with XLRS compared to fathers of sons with XLRS and a preliminary personality profile of mothers and fathers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants may be eligible to take part in this study if they: Have a biological son of any age with XLRS who is enrolled in XLRS Clinical and Molecular Studies protocol (03-EI-0033).

EXCLUSION CRITERIA:

-Participants may not be able to take part in this study if they:

* Are unable to understand and comply with the procedures of this study.
* Cannot communicate in English orally and in writing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 50 mothers of sons of all ages diagnosed with XLRS are eligible to participate in this study. Up to 50 fathers of sons of all ages with XLRS are also eligible to participate and will serve as a comparison group.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Description of the experiences of mothers of sons with XLRS compared to fathers of sons with XLRS | Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: Amy E Turriff, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States